CLINICAL TRIAL: NCT00569023
Title: Treatment of Congenital Stationary Night Blindness With an Alga Containing High Dose of Beta Carotene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ygal Rotenstreich, Opthalmologist, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-06-4496-YR-CTIL
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Night Blindness
Keywords: Beta Carotene; visual functions; Fundus albipunctatus; Night Blindness
MeSH Terms: conditions — Night Blindness; Fundus Albipunctatus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A,1,I (Experimental)
  Interventions: Dietary Supplement: alga Dunaliella bardawil

INTERVENTIONS:
Dietary Supplement: alga Dunaliella bardawil — Each patients will be treated with four capsules daily of Dunaliella bardawil for 90 days.
  Alga Dunaliella bardawil containing 15 mg approximately 50% all-trans beta-carotene and 50% 9-cis beta-carotene isomers

SUMMARY:
To assess the effect of oral administration of the alga Dunaliella bardawil containing approximately 50% all-trans beta-carotene and 50% 9-cis beta-carotene isomers on visual functions patients with Congenital Stationary Night Blindness {Fundus albipunctatus).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study.
* Men or women aged 18 years or older
* Diagnosed with Fundus albipunctatus

  1. Isolated rod response markedly reduced (less than 20% of normal)after 20 minutes dark adaptation and improved by 50% after 2 hours
  2. Negative maximal response (a wave to b wave ratio less than 2)
  3. Retinal midperipheral white dots (More than 3000 dots)

Exclusion Criteria:

* Current smokers.
* Current use of Vitamin A/ beta carotene supplements.
* Active arterial disease within 3 months of study entry such as unstable angina, myocardial infarction, transient ischemic attack (TIA), stroke, and coronary artery bypass graft (CABG) surgery.
* History of malignancy, except basal or squamous cell skin carcinoma.
* Pregnant women, women who are breast feeding, and women of childbearing potential who are not using chemical or mechanical contraception.
* Uncontrolled hypertension defined as either resting diastolic blood pressure of >95mmHg (taken from the mean of 3 readings) or resting systolic blood Pressure of > 180 mmHg.
* History of alcohol abuse or drug abuse, or both.
* Active liver disease or hepatic dysfunction as defined by elevations of 2.0 times the ULN in any of the following liver function tests: ALT, AST or bilirubin.
* Serum CPK > 2.0 times ULN in visit 0
* TSH above the normal range.
* Newly diagnosed diabetes within 3 months.
* Patient plans to engage in vigorous exercise or an aggressive diet regimen.
* Uncontrolled endocrine or metabolic disease.
* Participation in another investigational drug study within 4 weeks of entry into this study.
* Serious or unstable medical or psychological condition that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
* Serum creatinine > 2.0 mg/dl before the treatment phase, +3 proteinuria in urine dipstick, or a history of renal transplantation before the treatment period.
* Subject whose hormone replacement therapy (HRT) or oral contraceptive therapy (OCT) was initiated within the 3 month prior to enrollment.
* Forbidden medications: the combination of PPAR alpha agonists-fibric acid derivatives, PPAR gamma agonists.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-07; Primary Completion 2009-08 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Electroretinogram responses | Three months

SECONDARY OUTCOMES:
Visual acuity | Three Months

CONTACTS AND LOCATIONS:
Overall Officials: Ygal Rotenstreich, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel